CLINICAL TRIAL: NCT02832726
Title: TRIM: Danish Form and Dose Study in Vitamin B12
Brief Title: TRIM: Danish Form and Dose Study on Vitamin B12
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: KBA B48 2013
Record Dates: First submitted 2016-06-28; First posted 2016-07-14 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-06

CONDITIONS: Healthy
Keywords: absorption of Vitamin B12
MeSH Terms: interventions — Vitamin B 12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- cyano-hydroxo B12 (Active Comparator): Absorption of 3 doses of 9 ug cyano-B12 and 9 ug hydroxo-B12 for two days (the CobaSorb test). No drugs given.
  Interventions: Dietary Supplement: Vitamin B12
- Cyano-B12 doses (Active Comparator): Absorption of 3 doses of 3 ug, 6 ug, and 9 ug cyano-B12 for two days (the CobaSorb test). No drugs given.
  Interventions: Dietary Supplement: Vitamin B12

INTERVENTIONS:
Dietary Supplement: Vitamin B12
  Other Names: Cobalamin

SUMMARY:
The study investigates the absorption of different doses of hydroxocobalamin and cyanocobalamin in a vitamin B12-replete Danish population.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old

Exclusion Criteria:

* Use of vitamin pills with vitamin B12 within the last two weeks of the study
* Treatment with vitamin B12 injections within the last year
* Known chronic systemic disease
* Not able to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2014-01; Primary Completion 2016-05 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Vitamin B12 absorption (increase in holotranscobalamin) | 3 days

IPD SHARING:
Plan to Share IPD: No
No plan at this point

REFERENCES:
- [Derived] Greibe E, Mahalle N, Bhide V, Heegaard CW, Naik S, Nexo E. Increase in circulating holotranscobalamin after oral administration of cyanocobalamin or hydroxocobalamin in healthy adults with low and normal cobalamin status. Eur J Nutr. 2018 Dec;57(8):2847-2855. doi: 10.1007/s00394-017-1553-5. Epub 2017 Oct 16. PMID 29038891